CLINICAL TRIAL: NCT07237334
Title: A Prospective Cohort Study of the Clinical and Process Outcomes of Older Adults That Transition Through the Geriatric Emergency Medicine Unit (GEM-U)
Brief Title: A Prospective Cohort Study of Clinical and Process Outcomes of Older Adults That Transition Through the Geriatric Emergency Medicine Unit(GEM-U)
Status: Recruiting | Type: Observational
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Other Study IDs: GEM-U2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Frailty
Keywords: Comprehensive Geriatric Assessment
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will characterise the patients using the Geriatric Emergency Medicine Unit, a unit which provides specialist care for patients aged 75 years and older attending the emergency department. It will examine how this specialist care impacts their health in terms of a number of different outcomes, such as; function, quality of life and health care usage; for example admission to the acute hospital.

DETAILED DESCRIPTION:
The emergency department is a particularly challenging and busy environment, particularly for older adults living with frailty. It is widely acknowledged throughout the literature and national healthcare strategy that these older adults require holistic, person centred care that targets the intricacies of multifaceted, complex health issues.

The geriatric emergency medicine unit (GEM-U) aims to provide such care through the framework of comprehensive geriatric assessment, with in-put from a team of healthcare disciplines. The main aim of this study is to look at how this specialist care impacts patient outcomes, such as acute admission. Clinical and process outcomes of participants will be examined using patient reported outcome measures, which will include;

1. Global measure of function (Barthel Index)
2. Delirium screen (4AT +/- Delirium Rating Scale)*
3. Frailty status (Clinical Frailty Scale)
4. Nutritional status (Mini Nutritional Assesment)
5. Quality of life (EuroQoL-5D-5L).
6. Patient satisfaction (PSQ-18).

Participants will be followed at 30 days and 6 months post recruitment. All participants will give fully informed consent. The STrengthening the Reporting of OBservational studies in Epidemiology (STROBE) standardised reporting guidelines will be followed in the conduct and reporting of this research. Data will be statistically analysed

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged ≥75 years
* Manchester Triage System category 2-5
* Screen positive for risk of adverse outcomes after ED visit (≥ 2 on ISAR screening tool)
* Presenting with a medical condition
* Reviewed by the Older Persons Integrated Care Team

Exclusion Criteria:

* Patients presenting with a non-medical issue including major trauma or hip fracture

  * Patients presenting with acute stroke or transient ischaemic attack
  * Patients more appropriate to another alternative pathway e.g. deep vein thrombosis pathway, low risk chest pain pathway
  * Patients with acute coronary syndrome or unstable arrthymia
  * Patients requiring care in the resuscitation room
  * Patients with head injury (unless appropriate assessment and management has been fully completed by ED team)
  * Patients with possible spinal injury (unless appropriate assessment and management has been fully completed by ED/orthopaedic team)
  * Patients with low Glasgow Coma Scale
  * Other exclusions at the discretion of the Older Persons Integrated Care team depending on team capacity and expertise
  * Exclusion criteria as set out above, are in line with those set out in the UHL Operating Policy of the Older Persons Integrated Care Team.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All prospective older adults attending the GEMU that meet inclusion criteria will be invited to participate. However, this will be limited to the working hours of the research team (Monday-Friday, 8:00-20:00).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Our primary outcome is incidence of hospital admission at index GEM-U presentation | Patients are followed at 30 days and 6 months
  Patients who attend GEM-U and have an acute hospital admission at this time

SECONDARY OUTCOMES:
Mortality | Patients are followed at 30 days and 6 months
  Mortality
Unscheduled ED revisit | Patients are followed at 30 days and 6 months
  Patients who attend the ED department again during the follow up period
Unscheduled hospital visit(s) | Patients are followed at 30 days and 6 months
  Patients who have unplanned hospital admission (i.e. not elective procedure) during follow up period
Nursing home admission | Patients are followed at 30 days and 6 months
  Patients now living in a nursing home
Healthcare utilization (GP visit, out-patient geriatric services, PHN visit, HSCP services) | Patients are followed at 30 days and 6 months
  Use of primary care and community care services

CONTACTS AND LOCATIONS:
Overall Officials: Ida Carroll, Principal Investigator — University of Limerick
Locations (1):
- University Hospital Limerick, Limerick, Munster, Ireland